CLINICAL TRIAL: NCT04941157
Title: United States Aortic Research Consortium (ARC) Pilot Study: Prophylactic vs Therapeutic Cerebrospinal Fluid Drain Placement During Endovascular Thoracoabdominal Aortic Aneurysm Repair
Brief Title: Prophylactic vs Therapeutic Cerebrospinal Fluid Drain Placement During Endovascular Thoracoabdominal Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Massachusetts, Worcester (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Adam W Beck, Professor of Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-300006588
Record Dates: First submitted 2021-06-10; First posted 2021-06-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Ischemia
MeSH Terms: conditions — Spinal Cord Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic cerebrospinal fluid drain placement (Experimental): Patients randomized to receive the experimental treatment will have a prophylactic cerebrospinal fluid drain placed prior to their endovascular aortic repair. All components of the endovascular aortic repair are standard of care treatments.
  Interventions: Procedure: Cerebrospinal Fluid Drain Placement
- Selective cerebrospinal fluid drain placement (No Intervention): Patients randomized to the control arm of the study will not receive a prophylactic cerebrospinal fluid drain prior to their endovascular aortic repair. Patients will receive a CSF drain post-operative as needed to treat any symptoms of spinal cord ischemia. This arm of the study is current standard of care.

INTERVENTIONS:
Procedure: Cerebrospinal Fluid Drain Placement — Prophylactic CSF Spinal Drain to be placed prior to surgery in patients randomized to the experimental arm of the study
  Arms: Prophylactic cerebrospinal fluid drain placement

SUMMARY:
This is a pilot study to be performed at the University of Alabama at Birmingham (UAB) and the University of Massachusetts to determine the feasibility and develop the processes for a future randomized controlled trial to evaluate the occurrence of spinal cord ischemia after endovascular thoracoabdominal aneurysm repair using prophylactic cerebrospinal fluid drains versus no pre-emptive drain. The research question to be addressed is as follows: In the setting of a comprehensive spinal cord ischemia prevention protocol, do prophylactic CSF drains decrease the rate of spinal cord ischemia (SCI) in patients undergoing endovascular thoracoabdominal aneurysm repair?

DETAILED DESCRIPTION:
Endovascular techniques have transformed the management of thoracoabdominal (extending from the chest into the abdomen) aneurysms, with reduced early complications and death rates compared to open aortic repair operations.

However, injury to the spinal cord from reduced blood flow, termed spinal cord ischemia (SCI), continues to be a potentially devastating complication of these operations. SCI occurs in 2% to 15% of patients undergoing Thoracic and Thoracoabdominal Endovascular Aneurysm Repair, depending on length of aortic coverage, among other risk factors for SCI1. Paralysis and paraplegia resulting from SCI can be lead to profound long-term disability, as well as increased short and medium-term mortality. Only 25% of patients with permanent paralysis survive to one year due to complications that develop from SCI2. Additionally, SCI has tremendous financial consequences at many levels for the patient and the healthcare system, given the increased length of hospital/rehabilitation stay and the increased use of healthcare resources required for a paralyzed patient.

The avoidance of SCI is therefore critically important. Given the impact that SCI has on quality of life and survival after endovascular repair, avoidance of this complication is critical to the clinical success of the operation.

A number of strategies are in use to reduce the risk of developing SCI. These include elevation of the mean arterial pressure (blood pressure) to increase blood flow to the spinal cord, maintenance of an appropriate minimum hemoglobin concentration to improve oxygenation, prophylactic cerebrospinal fluid (CSF) drainage, as well as a number of procedural manipulations that are performed to decrease the occurrence of SCI3. CSF drainage is thought to improve spinal cord perfusion pressure by lowering the intraspinous pressure and thus increase the spinal cord perfusion pressure, given that the spinal cord perfusion pressure is the difference between mean arterial blood pressure and intraspinous pressure. Although prophylactic CSF drainage is widely used and conceptually attractive, it remains controversial due to its own inherent risk of complications4.

Despite its widespread use, the clinical effectiveness of prophylactic CSF drainage has not been definitively established, and the placement of these drains has a number of potential complications, including life threatening intracranial (brain) bleeding or spinal cord injury due to epidural (ie around the spinal cord) bleeding. There have been three randomized clinical trials of CSF drainage in patients undergoing open thoracoabdominal aortic surgery repair that demonstrated clinical effectiveness of CSF pressure drainage5. While these trials have some bearing on endovascular treatment, the findings are not fully generalizable to endovascular repairs given the inherent differences in the procedures and patient populations. Furthermore, these trials were conducted in the 1990s/early 2000s, and many aspects of perioperative care have changed since then, again limiting the applicability of the findings.

SCI has a spectrum of outcomes after it occurs, and may improve immediately with rescue maneuvers, or can lead to permanent paralysis. CSF drains can be placed prophylactically or placed post-operatively only if SCI develops6, which is often referred to as selective CSF drain placement. Prophylactic CSF drains have not been demonstrated to definitively prevent nor mitigate the severity of SCI in endovascular thoracoabdominal aortic repair, and it is not known whether outcomes of prophylactic drains are superior to selective drains7. Thus, many patients treated with prophylactic drains are put at risk for complications of drain placement and may not benefit from placement of the drain. Further, the strategies mentioned above for avoidance of SCI in the setting of potential CSF drain complications have lowered the incidence of SCI to a point where there is equipoise of prophylactic CSF drains versus selective drains, placed postoperatively only if SCI develops.

Demonstrative of this equipoise, standard of care is considered to be either prophylactic OR selective drain usage, depending on the surgeon and institution. Given this clinical equipoise, our intention is to evaluate the incidence of and outcomes of SCI with a pre-emptive CSF strategy versus placement only if SCI develops.

This is a pilot study to be performed at the University of Alabama at Birmingham (UAB) and the University of Massachusetts (UMass) to determine the feasibility and develop the processes for a future randomized controlled trial to evaluate the occurrence of SCI after endovascular thoracoabdominal aneurysm repair using prophylactic cerebrospinal fluid drains versus no pre-emptive drain. The research question to be addressed is as follows: In the setting of a comprehensive SCI prevention protocol, do prophylactic CSF drains decrease the rate of SCI in patients undergoing endovascular thoracoabdominal aneurysm repair?

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Undergoing high risk endovascular thoraco-abdominal aortic aneurysm repair, based on aortic coverage length:

2a: Extent I, II, III TAAA 2b: Extent IV TAAA with >5cm coverage above the celiac artery

Exclusion Criteria:

1. Active prison incarceration
2. active pregnancy
3. moribund patients
4. ruptured aneurysm
5. coagulopathy precluding CSF drain placement
6. urgent or emergent aneurysm repairs

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of Spinal Cord Ischemia Onset | Baseline to 1 year
  The primary outcome of this study is the rate of post-operative spinal cord ischemia. Onset of spinal cord ischemia will be defined by any new lower extremity neurologic deficit not attributable to another cause. Details of lower extremity neurologic exam will be collected during physical exam. Motor weakness will be measured using the Muscle Power Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Beck, MD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - Univeristy of Alabama at Birmingham Hospital, Birmingham, Alabama
  - UMass Memorial Health Hospital, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected electronically from UAB powerchart and stored in an encrypted and secure REDCap database (advanced clinical software application for data warehousing and healthcare analytics related to clinical trials) maintained centrally by UAB. Access to data will be limited to remembers of the research team identified on this IRB proposal. All shared data will be deidentified and related to procedural details and clinical outcomes. Data will be shared with the research team at the University of Massachusetts.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 month to 1 year
Access Criteria: Access to data will be limited to remembers of the research team identified on this IRB proposal.